CLINICAL TRIAL: NCT06734572
Title: 18F-FAPIBiotin PET/CT: Dosimetry and Biodistribution Study in Patients With Various Cancers
Brief Title: 18F-FAPIBiotin PET/CT: Dosimetry and Biodistribution Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-18F-FAPIBiotin
Record Dates: First submitted 2024-11-28; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dynamic PET scans (Experimental): PET imaging will begin at 3 minutes, 15 minutes, 30min minutes, 60 minutes and 120 minutes after injection.
  Interventions: Drug: 18F-FAPIBiotin

INTERVENTIONS:
Drug: 18F-FAPIBiotin — The dose will be 148-296 MBq given intravenously.

SUMMARY:
As a new dual targeting PET radiotracer, 18F-FAPI-Biotin is promising as an excellent imaging agent applicable to various cancers. In this study, we observed the safety, biodistribution and radiation dosimetry of 18F-FAPI-Biotin in patients with various types of cancer and compared them with the results of 18F-FAPI or 18F-FDG imaging to evaluate the dosimetric characteristics and diagnostic efficacy of 18F-FAPI.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is highly expressed in the stroma of a variety of human cancers and is therefore considered promising for guiding targeted therapy. The recent development of quinoline-based PET tracers that act as FAP inhibitors (FAPIs) demonstrated promising results preclinically and already in a few clinical cases. Biotin is overexpressed in various tumor cells and underexpressed in normal cells. We assume that expanding molecular probes targeting FAPI and biotin with dual targets to enhance the targeting ability of the tracer, improve the sensitivity and specificity of tumor lesion detection. 18F-FAPI-Biotin is a novel dual targeting tracer. The present study aimed to evaluate the biodistribution, pharmacokinetics, and dosimetry of 18F-FAPI-Biotin, and performed a head-to-head comparison with 18F-FAPI or 18F-FDG PET/CT scans in patients with various cancers.

ELIGIBILITY:
Inclusion Criteria:

* Various solid tumors with available histopathological findings • Signed informed consent

Exclusion Criteria:

* pregnant or lactational women • who suffered from severe hepatic and renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dosimetry of normal organs and tumors | From right after tracer injection to 120 minutes at post-injection
  The semiquantitative dosimetry will be performed based on PET/CT acquisitions after the first administration of 18F-FAPI-Biotin. The dose delivered to normal organs and tumors will be recorded.

SECONDARY OUTCOMES:
Incidence of Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0. | up to 1 week
  safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China